CLINICAL TRIAL: NCT04690907
Title: Dietary Intervention for Obese Pregnant Women - a Randomized Controlled Trial
Brief Title: Intervention, Dietary, Diabetes, Pregnancy
Acronym: IDDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Reeta Lamminpää, Post doctoral researcher, University of Eastern Finland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 031220
Record Dates: First submitted 2020-12-03; First posted 2020-12-31 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Dietary Habits; Obesity; Gestational Diabetes; Gestational Weight Gain
MeSH Terms: conditions — Feeding Behavior; Obesity; Diabetes, Gestational; Gestational Weight Gain | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Intervention group and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Dietary intervention: Written material on healthy diet during pregnancy, 2 virtual dietary counseling sessions given by a dietician. Otherwise basic care and counseling at maternity care clinics.
  Interventions: Behavioral: Dietary intervention
- Control group (No Intervention): Written material on healthy diet during pregnancy, otherwise basic care and counseling at maternity care clinics.

INTERVENTIONS:
Behavioral: Dietary intervention — Written material on healthy diet during pregnancy and 2 virtual dietary counseling sessions.
  Arms: Intervention group

SUMMARY:
The aim of this rct -study is to explore the effect of a dietary intervention for overweight (body maas index BMI≥25) and obese (BMI≥30) pregnant women on gestational weight gain and the prevalence of gestational diabetes.

DETAILED DESCRIPTION:
Pregnant women are recruited for the study from 18 maternity care clinics in Northern Savo and Northern Karelia area. The participants will be randomized into intervention and control groups. All the participants will have access to the study web-pages, which includes written material of healthy diet during pregnancy as well as all the study material (4 day food records, Three factor eating questionnaire (TFEQ R-18) and Binge Eating Scale (BES)). In addition, intervention group will get two virtual dietary counseling sessions by a dietician. The information on participants' gestational weight gain and the result of oral glucose tolerance tests will be collected by the public health nurses after birth.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25 or higher
* healthy, no chronic medical conditions that can prevent participating to the study
* singleton pregnancy
* first trimester of pregnancy at the time of recruitment

Exclusion Criteria:

* BMI less than 25
* chronic medical conditions
* multiple pregnancy
* pregnancy at second or third trimester at the time of recruitment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females because of pregnancy
Enrollment: 33 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain (GWG) | immediately after the intervention
  gestational weight gain (from pre-pregnancy weight until childbirth), measured at maternity care clinic.

SECONDARY OUTCOMES:
Gestational diabetes mellitus (GDM) | immediately after the intervention
  GDM is measured by the result of an oral glucose tolerance test (OGTT)
Eating habits I | During the intervention up to gestational weeks 36-37
  eating habits are measured by 4 day food records
Eating habits II | During the intervention up to gestational weeks 37-42
  Eating habits are measured by TFEQ R-18 questionnaire
Eating habits III | During the intervention up to gestational weeks 37-42
  Eating habits are measured by Binge Eating Scale (BES)

CONTACTS AND LOCATIONS:
Overall Officials: Reeta Lamminpää, Principal Investigator — University of Eastern Finland
Locations (2):
- Finland (2):
  - Antenatal maternity care clinics (n=6), Joensuu
  - Antenatal maternity care clinics (n=12), Kuopio

IPD SHARING:
Plan to Share IPD: No